CLINICAL TRIAL: NCT03086304
Title: Effects of Transcutaneous Acupoint Electrical Stimulation on Intestinal Obstruction After Gastrointestinal Surgery in Adults
Brief Title: Effects of Transcutaneous Acupoint Electrical Stimulation on Intestinal Obstruction After Gastrointestinal Surgery
Acronym: TAESRIOGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Shaanxi Provincial People's Hospital (Other); Xi'an Central Hospital (Other); Ankang Hospital of Traditional Chinese Medicine (Other); Affiliated Hospital of Shaanxi University of traditional Chinese Medicine (Unknown); Ankang Central Hospital (Other); Weinan Central Hospital (Other); Central Railway Group of Xi'an Central Hospital (Unknown); Xi'an Hospital of Traditional Chinese Medicine (Other); Yan'an University Affiliated Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2016-003
Record Dates: First submitted 2017-03-03; First posted 2017-03-22 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Intestinal Obstruction
Keywords: postoperative intestinal obstruction;TEAS

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAS group (Experimental): Choose several acupoints,give 2/10 hz dilatational wave stimulation.Complete the 30 minutes intervention after extubation and 1-3 days after surgery.Give a health education on the first postoperative day.
  Interventions: Device: transcutaneous acupoint electrical stimulation
- no TEAS group (Experimental): The choice of acupoints are same with TEAS group,tape over the electrode but don't give electroacupuncture stimulation,the others steps are same with TEAS group.
  Interventions: Device: no transcutaneous acupoint electrical stimulation

INTERVENTIONS:
Device: transcutaneous acupoint electrical stimulation — Transcutaneous acupoint electrical stimulation is same to the traditional Chinese medicine acupuncture treatment,treat diseases by stimulate different acupuncture points.
  Arms: TEAS group
Device: no transcutaneous acupoint electrical stimulation — the choice of acupoints are same with TEAS group,tape over the electrode but don't give electroacupuncture stimulation.
  Arms: no TEAS group

SUMMARY:
Postoperative intestinal obstruction (POI) is one of the most common complications in the gastrointestinal surgery. Compared with the conventional control group, transcutaneous acupoint electrical stimulation(TEAS) is possible to reduce the incidence of POI and accelerate the rapid recovery of the gastrointestinal tract.

DETAILED DESCRIPTION:
Participants will be randomly assigned, in a 1:1 ratio, to receive TEAS or Blank treatment (acupoints selection are same with the experimental group, connect stimulator for patients, but not don't give stimulus). The randomization sequence will be computer-generated, and randomization will be performed in blocks and will be stratified according to participating center. TEAS will be performed in a series of time periods after operation. Time of first fart and food-taking ,time of have normal diet after the transplantation will be recorded. The participation of each patient is scheduled for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* All the patients signed the informed consent before treatment;
* Age ≥ 18 years old,American society of Anesthesiologists(ASA)grade are between I and III;
* Plan to perform elective colon and rectal tumor resection under general anesthesia;
* not involved in other clinical studies;
* no cognitive impairment, mental disorders,communication disorders.

Exclusion Criteria:

* Pregnancy, breast-feeding;
* The history of intestinal surgery;
* Test point skin injury, infection, allergies to tape;
* have undergone external enterostomy;
* Chief surgeon refuse to cooperate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of POI | 72 hours after surgery
  Whether or not to exhaust in 72 hours after surgery

SECONDARY OUTCOMES:
postoperative gastrointestinal function recovery | once a week for 30 days after surgery
  the time of postoperative exhaustion and defecation.
recovery of bowel sounds | 1-3 days after surgery
  the recovery time of bowel sounds
adverse reactions of digestive after surgery | 1-3 days after surgery
  the incidence and score of distention, abdominal pain, nausea and vomiting after surgery.
surgery complications | once a week for 30 days after surgery
  wound infection ,pneumonia, anastomotic leakage,urethritis,uroschesis
recovery index | once a week for 30 days after surgery
  the leaving bed time,normal diet recovery time,post-operative hospitalization duration

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, PHD, Study Chair — First Affiliated Hospital of Xian JiaotongUniversity
Locations (10):
- China (10):
  - Ankang Central Hospital, Ankang, Shaanxi
  - Ankang Hospital of Traditional Chinese Medicine, Ankang, Shaanxi
  - Weinan Central Hospital, Weinan, Shaanxi
  - Xi'an Central Hospital, Xi'an, Shaanxi
  - Xi'an Hospital of traditional Chinese Medicine, Xi'an, Shaanxi
  - Central Railway Group of Xi'an Central Hospital, Xi'an, Shaanxi
  - First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Affiliated Hospital of Shaanxi University of traditional Chinese Medicine, Xianyang, Shaanxi
  - Affiliated Hospital of Yan'an University, Yan’an, Shaanxi

IPD SHARING:
Plan to Share IPD: Undecided